CLINICAL TRIAL: NCT04733066
Title: Quality of Life in Patients With Short Bowel Syndrome Treated Without and With Teduglutide - a Prospective Nested Matched Pair Analysis
Acronym: MatchedQoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Elisabeth Blüthner, MD, Charite University, Berlin, Germany
Other Study IDs: IIR-DE-002726
Record Dates: First submitted 2020-08-29; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Short Bowel Syndrome; Intestinal Failure
Keywords: Quality of Life; Teduglutide; GLP-2 Analogue
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure | interventions — teduglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-treatment Group: 1. Quality of life assessment (SBS-QoL, SF- 36)
  2. Nutrition status assessment (BIA, BMI)
  3. Assessment of functional absorptive small bowel length (citrulline)
  4. Clinical data (nutritional program, stool characteristics)
- Teduglutide-treated Group: 1. Quality of life assessment (SBS-QoL, SF- 36)
  2. Nutrition status assessment (BIA, BMI)
  3. Assessment of functional absorptive small bowel length (citrulline)
  4. Clinical data (nutritional program, stool characteristics)
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Intervention group consists of patients, who receive teduglutide within routine medical care
  Groups: Teduglutide-treated Group

SUMMARY:
The aim of this prospective longitudinal study is to compare the quality of life of short bowel patients prior to and on teduglutide treatment with a non-treated patient group in a matched-pair design.

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is a malabsorptive disorder mostly caused by surgical interventions, which may result in chronic intestinal failure (cIF). The incidence is progressively increasing due to more aggressive surgical and medical approaches. Parenteral nutrition is still the mainstay of treatment for patients with irreversible cIF. New hormonal therapies hold promise by romoting mucosal growth and intestinal absorption and thereby leading to a consequent reduction in parenteral support and symptoms related to large stomal or faecal losses. Outside the typical primary endpoints of cost data, quality of life (QoL) is an important and yet underappreciated consideration of the effectiveness of targeted therapies. In the clinical STEPS trial, Jeppesen et al. have previously shown a significant improvement of the SBS-QoL total score after 24 week treatment with teduglutide longitudinally but could not identify a statistical significance to the placebo group. Accordingly, Chen and colleagues carried out a post hoc analysis of the afore mentioned clinical trial data based on 86 patients and could confirm the results auf Jeppesen et al. Taken together, these clinical trial data did not show a direct benefit of teduglutide treatment on QoL in these patients, while real life data on QoL changes are not available yet. During the release of teduglutide in Germany, the PNLiver trial (DRKS00010993) recruited chronic intestinal failure patients with parenteral nutrition from 2014 till 2019 to evaluate the capability of non-invasive liver function tests in cIF patients in a cross-sectional (n=90) and longitudinal study (n=20. All participants underwent study visits including clinical examination, dynamic liver function assessment, comprehensive blood tests, nutritional status assessment and quality of life assessment (Short Form 36 [SF-36] and SBS-QoL). Therefore, we have a comprehensive data set of a large monocentric cIF cohort prior to teduglutide treatment. Consequently, our unique QoL data from the PNLiver trail enables a followup assessment for an observation period above 24 weeks of patients who were in the meantime exposed to teduglutide in a real life setting. Nevertheless, QoL also tends to improve with longer duration on HPN. Therefore, we are aiming to extend the results with a pairwise matched control group from non teduglutide-treated PNLiver trail patients and collect follow-up data from this group accordingly.

ELIGIBILITY:
Inclusion Criteria:

* SBS-associated adult chronic IF with parenteral nutritional support
* previous inclusion in the PNLiver trial with existing SF-36 and SBSQoL data
* signed informed consent

Exclusion Criteria:

* teduglutide stop before study initiation
* refusal or withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A comprehensive data set of a large monocentric cIF cohort prior to teduglutide treatment from the PNLiver trail already exists. Consequently, we aim to have a follow-up assessment of patients who are in the meantime treated with teduglutide as a clinical routine procedure.
  We aim to extent the results with a pairwise matched control group from non teduglutide-treated PNLiver trail patients and collect follow-up data from this group accordingly.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
changes in QoL data during teduglutide therapy | through study completion, an average of 1 year
  SBS-QoL, SF-36
changes in QoL data of patients without teduglutide therapy | through study completion, an average of 1 year
  SBS-QoL, SF-36
changes in QoL data of teduglutide treated patients compared to changes in pairwise matched controls | through study completion, an average of 1 year
  SBS-QoL, SF-36

SECONDARY OUTCOMES:
BMI in kg/m^2 | through study completion, an average of 1 year
  weight and height will be combined to report BMI in kg/m^2
Body cell mass in kg | through study completion, an average of 1 year
  measured by bioelectrical impedance analysis
citrulline levels | through study completion, an average of 1 year
stool characteristics by bristol stool scale | through study completion, an average of 1 year
  seven types of stool from 1 (hard lumps) till 7 (watery)
parenteral support frequency | through study completion, an average of 1 year
parenteral support volume | through study completion, an average of 1 year
parenteral support calories | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeppesen PB, Pertkiewicz M, Forbes A, Pironi L, Gabe SM, Joly F, Messing B, Loth S, Youssef NN, Heinze H, Berghofer P. Quality of life in patients with short bowel syndrome treated with the new glucagon-like peptide-2 analogue teduglutide--analyses from a randomised, placebo-controlled study. Clin Nutr. 2013 Oct;32(5):713-21. doi: 10.1016/j.clnu.2013.03.016. Epub 2013 Mar 28. PMID 23587733
- [Background] Chen K, Mu F, Xie J, Kelkar SS, Olivier C, Signorovitch J, Jeppesen PB. Impact of Teduglutide on Quality of Life Among Patients With Short Bowel Syndrome and Intestinal Failure. JPEN J Parenter Enteral Nutr. 2020 Jan;44(1):119-128. doi: 10.1002/jpen.1588. Epub 2019 Apr 21. PMID 31006876
- [Background] Bluthner E, Bednarsch J, Pape UF, Karber M, Maasberg S, Gerlach UA, Pascher A, Wiedenmann B, Pratschke J, Stockmann M. Advanced liver function assessment in patients with intestinal failure on long-term parenteral nutrition. Clin Nutr. 2020 Feb;39(2):540-547. doi: 10.1016/j.clnu.2019.02.039. Epub 2019 Mar 5. PMID 30885502
- [Background] Bluthner E, Bednarsch J, Stockmann M, Karber M, Pevny S, Maasberg S, Gerlach UA, Pascher A, Wiedenmann B, Pratschke J, Pape UF. Determinants of Quality of Life in Patients With Intestinal Failure Receiving Long-Term Parenteral Nutrition Using the SF-36 Questionnaire: A German Single-Center Prospective Observational Study. JPEN J Parenter Enteral Nutr. 2020 Feb;44(2):291-300. doi: 10.1002/jpen.1531. Epub 2019 Mar 13. PMID 30864177